CLINICAL TRIAL: NCT05866627
Title: A Phase 1 Open-label, 2-Part Crossover Study to Assess the Effect of Acid-reducing Agent Famotidine on the Pharmacokinetics of Afimetoran (BMS-986256) in Healthy Participants
Brief Title: A Study to Assess the Effect of Famotidine on the Drug Levels of Afimetoran in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM026-1023; 1007296 (Other: IRAS)
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers
Keywords: BMS-986256; Famotidine; Gastric pH
MeSH Terms: interventions — Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Afimetoran, followed by famotidine + afimetoran (Experimental)
  Interventions: Drug: Famotidine; Drug: Afimetoran
- Famotidine + afimetoran, followed by afimetoran (Experimental)
  Interventions: Drug: Famotidine; Drug: Afimetoran
- Afimetoran (Experimental)
  Interventions: Drug: Afimetoran
- Famotidine, followed by afimetoran (Experimental)
  Interventions: Drug: Famotidine; Drug: Afimetoran

INTERVENTIONS:
Drug: Famotidine — Specified dose on specified days
  Other Names: Pepcid
  Arms: Afimetoran, followed by famotidine + afimetoran; Famotidine + afimetoran, followed by afimetoran; Famotidine, followed by afimetoran
Drug: Afimetoran — Specified dose on specified days
  Other Names: BMS-986256

SUMMARY:
The purpose of this study is to confirm there is no significant effect of gastric pH changes of famotidine on the drug levels of afimetoran in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥ 50 kilograms (kg), at screening and first admission, and body mass index between 18.0 kilogram per square meter (kg/m^2) and 32.0 kg/m^2, inclusive, at screening.
* A negative QuantiFERON-TB Gold test result at screening or documentation of a negative result within 3 months before screening.
* Normal renal function at screening as evidenced by an estimated glomerular filtration rate (eGFR) ≥ 80 milliliter per minute (mL/min)/1.732 m^2 calculated with the Chronic Kidney Disease Epidemiology Collaboration formula.

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Current or recent (within 3 months of study drug administration) gastrointestinal (GI) disease that could impact upon the absorption of study treatment.
* GI surgery, including cholecystectomy, that could impact upon the absorption of study treatment, at the investigator's discretion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 20 Days
Time to attain maximum observed plasma concentration (Tmax) | Up to 20 Days
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration (AUC[0-T]) | Up to 20 Days

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 52 Days
Number of participants with clinical laboratory abnormalities | Up to 52 Days
Number of participants with vital sign abnormalities | Up to 52 Days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 52 Days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Quotient Sciences, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com